CLINICAL TRIAL: NCT00076284
Title: A Phase II, Double-Blind RAndomized, Placebo-Controlled Study to Evaluate the Antiviral Activity, Safety, Tolerability, and Pharmacokinetics of GW873130 for 10 Days in HIV-1 Infected Adults
Brief Title: GW873140 to Treat HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040087; 04-I-0087
Record Dates: First submitted 2004-01-16; First posted 2004-01-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: HIV Infections
Keywords: CCR5 Antagonist; Coreceptor Inhibitor; Fusion Inhibitor; Entry Inhibitor; Antiretroviral; HIV
MeSH Terms: conditions — HIV Infections | interventions — aplaviroc

INTERVENTIONS:
Drug: GW873140

SUMMARY:
This study will determine which of four doses of GW873140 can safely be given to adults to lower the amount of virus (HIV-1) in the body. GW873140 is a new type of anti-HIV drug called a CCR5 receptor antagonist. CCR5 is a receptor on T cells (a type of white blood cell) where HIV-1 enters and then infects the cell. GW873140 is intended to block the CCR5 receptor so that HIV-1 cannot enter the cell.

HIV-1-infected patients 18 years of age and older may be eligible for this study. Candidates are screened with a medical history and physical examination, electrocardiogram, and blood and urine tests. Some of the blood drawn is used to test the patient's HIV-1 type to see if the study drug might lower the amount of HIV-1 in the blood. Women who can become pregnant have a pregnancy test.

Participants are hospitalized for 12 days. They are randomly assigned to take one of the following four treatments for 10 days: 1) 200 mg of GW873140 once a day, or placebo (a look-alike pill with no active ingredient); 2) 200 mg of GW873140 twice a day, or placebo; 3) 400 mg of GW873140 once a day, or placebo; or 600 mg of GW873140 twice a day, or placebo. Participants record the meals they eat on a diary card. In addition, they undergo the following tests and procedures:

During treatment

* Assessment of HIV classification (day 1)
* Review of meal diary cards (days 1,2,3,4,5,8, and 10)
* Review of any HIV-associated conditions, other medications taken besides the study drug, and well-being (days 1,2,3,4,5,8,10, and 11)
* Check of vital signs, including blood pressure, pulse, and temperature (days 1,2,3,4,5,6,7,8,10, and 11)
* Weight assessment (days 1 and 10)
* Electrocardiogram to measure the electrical activity of the heart (days 1,2,3,8, and 10)
* Blood draws for routine laboratory tests, to measure T-cell counts, and to measure HIV levels (days 1,2,5,10, and 11)
* Urine tests (days 1 and 10)

Post-treatment

* Blood tests to monitor the effect of GW873140 on lowering HIV counts (days 12, 15, 17, and 19)

Follow-up visit (2 weeks after last drug dose--day 24)

* Review of medications taken and general well-being
* Check of vital signs
* Physical examination
* Blood and urine tests.

DETAILED DESCRIPTION:
The development of resistance to all currently marketed drugs for HIV infection has been observed and is a major reason for failure of therapy. In particular, there is a great need for drugs against new targets and having novel mechanisms of action against new targets. Most of the currently approved drugs are targeted toward the inhibition of viral enzymes. However, the process of viral entry and fusion has become an active area of research. Among the steps involved in viral entry, binding of HIV to CD4 co-receptors on the cell surface is an important and promising target for new drug development.

GW873140 is a CCR5 antagonist that is in Phase I clinical development as a viral entry inhibitor for the treatment of HIV infection. GW873140 has demonstrated in vitro antiviral activity with an IC50 against CCR5-tropic HIV-1 of 1nM equals about 0.5ng/mL), that is shifted 8-10 fold (10nM equals about 0.5ng/mL) in the presence of physiological concentrations of human plasma proteins. A study to investigate the safety, tolerability, and pharmacokinetics of escalating single (50-1200mg) and repeat (200-800mg BID) doses of GW873140 has been conducted in 70 healthy volunteers (GW873140/001). Preliminary results indicate that GW873140 is well-tolerated up to a dose of 1200 mg following single dose and 800 mg BID following multiple-dose. Additionally, food was shown to increase the AUC and Cmax of a 400 mg single dose by 1.7-and 2.2-fold, respectively.

Concentrations above the protein binding corrected IC90 are achieved following oral dosing and in vivo binding studies in healthy subjects demonstrate greater than 97% receptor occupancy 2 and 12 hours after multiple doses and 68-88% receptor occupancy 24 hours after a single dose, despite plasma concentrations below or near detectable limits.

ELIGIBILITY:
INCLUSION CRITERIA:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Healthy adult male aged greater than or equal to 18 OR

   Healthy adult female aged greater than or equal to 18, of non-childbearing potential, defined as: Women who are surgically sterile or are post-menopausal, as indicated by history of no menses for a minimum of one year from the date of the screening visit.

   Healthy adult female aged greater than or equal to 18 of childbearing potential, who agrees to use double barrier method (e.g. condom+diaphragm) starting from the screening visit through the follow up visit (Day 24).

   Note: Spermicides and/or hormonal contraceptives will not be considered sufficient forms of contraception for this study.
2. Screening plasma HIV-1 RNA greater than or equal to 5,000- less than or equal to 250,000 copies/mL.
3. Viral load within the past 30-90 days of the screening visit must be within 0.5log of screening HIV-1 RNA.
4. Not taken any antiretroviral therapy for the preceding 3 months from screening visit.
5. CD4 cell count greater than or equal to 200 cells/mm(3) with a historical nadir greater than or equal to 200 cells/mm(3).
6. CCR5-tropic virus based on viral tropism assessment at screening visit.
7. Normal resting 12-lead electrocardiogram at screening visit.
8. Signed and dated written informed consent prior to admission to the study.
9. In addition to the inclusion criteria listed above, patients must meet the following inclusion criteria:

   * Willingness and ability to fast for 10 hours except for water from 9:00 p.m. until 7:00 a.m. during eight of the study days.
   * Willingness and ability to eat a 30% fat diet during the 10 day treatment period of the study.
   * Willingness to allow stored blood samples to be used in the future for further testing or for studying HIV disease and immune function.

EXCLUSION CRITERIA:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. CXCR4 tropic virus based on viral tropsin assessment at screening visit.
2. Chronic diarrhea (greater than 3 stools/day)
3. Subject with history of oropharyngeal candidiasis or C AIDS-defining illness according to the 1993 Centers for Disease Control (CDC) AIDS surveillance definition.
4. Greater than two prior ARV regimens.
5. Any acute laboratory abnormality at screen which, in the opinion of the investigator, should preclude the subject's participation in the study of an investigational compound. Any grade 4 laboratory abnormality at screen will exclude a subject from study participation unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor.
6. Significant blood loss (1 pint of whole blood) within 56 days of the screening visit of the study.
7. Previous participation in an experimental drug trial(s) within 30 days of the screening visit of the study.
8. Any conduction delay, regardless of clinical significance on screening ECG.
9. History of clinically relevant pancreatitis or hepatitis within the previous 6 months.
10. Any condition which, in the opinion of the investigator, may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations (including alcohol or drug abuse) or which might compromise the safety of the subject.
11. Any condition which, in the opinion of the investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug such as diabetes mellitus, hyperthyroidism, malabsorption syndrome, etc.
12. History of cholecystectomy, cholelithiasis or cholecystitis.
13. Any immunization within 30 days prior to first dose of investigational product.
14. History of a drug or other allergy which in the opinion of the investigator, contraindicates the subject's participation in the study or known hypersensitivity to any study medication.
15. Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of investigational product administration or anticipated need for such treatment within the study.
16. Treatment with immunomodulating agents (such as interleukins, interferons) or any agents with known anti-HIV activity (such as hydroxyurea, foscarnet, or NRTIs) within 30 days of investigational product administration.
17. Use of steroids (oral) within 30 days of first dose of investigational product.
18. Prior treatment with any entry, attachment or fusion inhibitor, experimental or approved.
19. Pregnant women or women who are breastfeeding.
20. Subjects who cannot refrain from drinking grapefruit juice or eating grapefruit within 3 days prior to the first dose of study medication until collection of the final pharmacokinetic blood sample.
21. Use of prescription or non-prescription medications that are not on the GSK APPROVED MEDICATION LIST for GW873140.

Medications that are not approved on this list, will need to be discontinued 7 days prior to first dose of investigational product (for drugs that are non-hepatic inducers) and 30 days prior to first dose of investigational product (for drugs that are hepatic inducers) through 5 days post dose.

To clarify the exclusion of patients with hepatitis and pancreatitis, the following patients will be excluded:

* Patients with a diagnosis of acute viral hepatitis infection in the preceding six months
* Patients with a history of AST or ALT elevation five times normal or greater in the the preceding six months
* Patients who have been diagnosed with pancreatitis in the preceding six months or have had an elevation of lipase two times normal or greater and symptoms suggestive of pancreatitis (i.e. nausea, vomiting, epigastric pain).

Patients with evidence of chronic hepatitis B or C are not excluded from study participation if they are clinically asymptomatic, liver enzymes are less than five times normal, and they have no evidence of hepatic synthetic dysfunction (i.e. PT less than 1.5 times upper limit of normal).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-01; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Arranz M, Collier D, Sodhi M, Ball D, Roberts G, Price J, Sham P, Kerwin R. Association between clozapine response and allelic variation in 5-HT2A receptor gene. Lancet. 1995 Jul 29;346(8970):281-2. doi: 10.1016/s0140-6736(95)92168-0. PMID 7630250
- [Background] Blanpain C, Lee B, Tackoen M, Puffer B, Boom A, Libert F, Sharron M, Wittamer V, Vassart G, Doms RW, Parmentier M. Multiple nonfunctional alleles of CCR5 are frequent in various human populations. Blood. 2000 Sep 1;96(5):1638-45. PMID 10961858
- [Background] Cardon LR, Idury RM, Harris TJ, Witte JS, Elston RC. Testing drug response in the presence of genetic information: sampling issues for clinical trials. Pharmacogenetics. 2000 Aug;10(6):503-10. doi: 10.1097/00008571-200008000-00003. PMID 10975604